CLINICAL TRIAL: NCT04734158
Title: EVALUATION OF CORNEAL EPITHELIAL THICKNESS MAPPING IN DIABETIC PATIENTS USING ANTERIOR SEGMENT OPTICAL COHERENCE TOMOGRAPHY AND ITS CORRELATION TO MACULAR THICKNESS
Brief Title: CORNEAL EPITHELIAL MAPPING IN DIABETICS
Status: Active, not recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hosny Ahmed Zein, DR. HOSNY AHMED ZEIN, Minia University
Other Study IDs: MiniaUN
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Cornea Epithelial Mapping
Keywords: cornea epithelium OCT diabetes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control
  Interventions: Other: corneal imaging
- Diabetics with macular edema
  Interventions: Other: corneal imaging
- Diabetics without macular edema
  Interventions: Other: corneal imaging

INTERVENTIONS:
Other: corneal imaging — corneal imaging using AS-OCT

SUMMARY:
The corneal epithelium is the outermost layer that covers the front of the eye; it not only functions as a barrier that blocks the passage of foreign material, but also plays an important role in maintaining high optical quality. The stem cells in the basal layer of the limbal epithelium hold a physiological significance in the renewal and metabolism of corneal epithelium, particularly under stressful situations.

DETAILED DESCRIPTION:
The cornea in diabetic patients suffers from cellular dysfunction and dysfunctional repairal mechanisms, which include recurrent erosions, delayed wound healing, ulcers, and edema. In addition and undoubtedly related to epithelial dysfunction, alterations in epithelial basement membrane occur.

ELIGIBILITY:
Inclusion Criteria:

1. The patients aged between 40- 60 years old of both genders.
2. The patients in (Group A) should be diabetics for more than 10 years and free from any other systemic diseases with diabetic macular edema (by OCT).
3. The patients in (Group B) should be diabetics for more than 10 years and free from any other systemic diseases without diabetic macular edema (by OCT).
4. The patients in (Group C) should be free of any systemic diseases and normal macular thickness (by OCT)

Exclusion Criteria:

1. Previous history of any intraocular surgery, intravitreal injection, laser or refractive surgery.
2. Ocular surface disorders (e.g. dry eye) or any corneal pathology.
3. Corneal scars or epithelial dystrophies.
4. Use of any topical medications.
5. Elevated IOP, pregnancy or lactation.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It's a prospective cross section study. 159 eyes of 159 patients will be involved in this study, divided into three groups: (Group A) 53 eyes of diabetic patients with diabetic macular edema, (Group B) 53 eyes of diabetic patients without macular edema and (group C) 53 eyes of age matched control.
Sampling Method: Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
corneal epithelial thickness | 2 years
  corneal thickness in diabetics using OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided